CLINICAL TRIAL: NCT03220698
Title: Utility of Tracheal Ultrasonography for the Confirmation of Endotracheal Tube Placement During Intubation: A Diagnostic Accuracy Study
Brief Title: Utility of Tracheal Ultrasonography for the Confirmation of the Endotracheal Tube Placement
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Haldun Akoglu, Associate Professor of Emergency Medicine, Marmara University
Other Study IDs: 09.2016.054
Record Dates: First submitted 2017-07-14; First posted 2017-07-18 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Intubation Complication
Keywords: endotracheal intubation; confirmation; ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Tracheal ultrasonography — Tracheal ultrasonography

SUMMARY:
The aim of this study is to compare tracheal ultrasound with direct visualization of tracheal rings for the confirmation of endotracheal tube placement in intubated patients. We hypothesize that this method is more reliable, cheap, and readily available for all emergency physicians.

DETAILED DESCRIPTION:
Confirmation of the ETT placement has utmost importance in the management of airway in emergency medicine (EM). Visual examination of the tube (fogging), auscultation, chest x-ray, capnography, capnometry and fiberoptic bronchoscopy are the main tools used for confirmation with increasing diagnostic utilities. Recently, tracheal ultrasonography (US) was introduced as a reliable, cheap and readily available method of confirmation of ETT placement.

ELIGIBILITY:
Inclusion Criteria:

* adults (>=18 years)
* intubated in the ED
* during the shifts of the researchers (TM, OFC).

Exclusion Criteria:

* anatomical, traumatic or tumoral defect(s) at the site of sonographic imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible for the inclusion were consecutive adults (>=18 years) intubated in the ED during the shifts of the researchers (TM, OFC). We excluded patients if they have anatomical, traumatic or tumoral defect(s) at the site of sonographic imaging.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Presence of endotracheal tube in trachea | Immediately after the intubation process
  Whether the endotracheal tube is in the trachea or not

CONTACTS AND LOCATIONS:
Overall Officials: Haldun Akoglu, MD, Principal Investigator — Marmara University

IPD SHARING:
Plan to Share IPD: No